CLINICAL TRIAL: NCT06400784
Title: The Evidence-based Treatment of Hypertensive Heart Failure in Sub-Saharan Africa: A Feasibility Study
Brief Title: Hypertensive Heart Failure Treatment in SSA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Abuja (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Dr. Dike Ojji, Associate Professor, University of Abuja
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uniabuja; G 102642 A18971 (Other: University of Cambridge_GCFR)
Record Dates: First submitted 2022-12-31; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: A Feasibility Study on Hypertensive Heart Failure Treatment
MeSH Terms: interventions — Isosorbide Dinitrate

STUDY DESIGN:
Intervention Model Description: Parallel group, 2-arm, superiority trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional HF medications plus ISDN & HYD (Active Comparator): Will administer Isosorbide dinitrate (5mg bd) and Hydralazine (25mg bd) on top of conventional heart failure medications.
  Interventions: Drug: Isosorbide Dinitrate
- Conventional HF medications plus placebo (Placebo Comparator): We will administer placebo on top of conventional heart failure medications
  Interventions: Drug: Isosorbide Dinitrate

INTERVENTIONS:
Drug: Isosorbide Dinitrate — Isosorbide dinitrate (5mg bd) and Hydralazine (25mg bd) will be added on top of conventional heart failure medications.

SUMMARY:
Even though, the African-American Heart Failure Trial (A- HeFT) demonstrated that a combination ISDN and HYD (BiDil) improved survival among African-American patients with HF, when compared to placebo, there is no trial on chronic heart failure patients secondary to hypertensive heart disease which is the commonest etiological factor for heart failure in sub-Saharan Africa.

A previous study (The Bi treatment with hydralazine/nitrate versus placebo in Africans admitted with acute Heart Failure (BAHEF) which was on acute heart failure patients with varying aetiology, was under powered as the study could not achieve the estimated sample size because of logistic issues.

We therefore are trying to determine the feasibility of a randomised, open-label, parallel group, two-arm, superiority trial of ISDN and hydralazine in patients with chronic hypertensive heart failure in sSA.

DETAILED DESCRIPTION:
Even though, the African-American Heart Failure Trial (A- HeFT) demonstrated that a combination ISDN and HYD (BiDil) improved survival among African-American patients with HF, when compared to placebo, there is no trial on chronic heart failure patients secondary to hypertensive heart disease which is the commonest etiological factor for heart failure in sub-Saharan Africa.

A previous study (The Bi treatment with hydralazine/nitrate versus placebo in Africans admitted with acute Heart Failure (BAHEF) which was on acute heart failure patients with varying aetiology, was under powered as the study could not achieve the estimated sample size because of logistic issues.

We therefore are trying to determine the feasibility of a randomised, open-label, parallel group, two-arm, superiority trial of ISDN and hydralazine in patients with chronic hypertensive heart failure in sSA. To determine the tolerability of ISDN and hydralazine in sSA.

The secondary objectives on the other hand are:

1. To determine fidelity to the trial protocol and CRF by investigators when completing a trial utilising ISDN and hydralazine in patients with chronic hypertensive heart failure in sSA.
2. To determine the effect of ISDN-HYD on the following:

   * Death and hospitalisation rates
   * Changes in office BP
   * Changes in 6MWT
   * Changes in echocardiographic left ventricular ejection fraction

ELIGIBILITY:
Inclusion Criteria:

* Black male or female aged 18 years
* Evidence of hypertensive heart failure
* LVEF <40% as assessed by 2D echocardiography (modified Simpson method)
* Ability to provide written informed consent for participation in the study
* Available for regular follow-up as outlined in the schedule of assessments

Exclusion Criteria:

* Evidence of heart failure from a cause other than hypertension
* A cardiovascular/cerebrovascular event/intervention in the last three months (e.g., acute
* coronary syndrome, unstable angina, MI, PCI, CABG, stroke, carotid endarterectomy, etc.,)
* Office SBP <100 mmHg or DBP <70 mmHg
* Marked renal impairment (e.g., eGFR <45 mls/min at screening, dialysis)
* Marked hepatic impairment (e.g., history of chronic liver disease, γGT/bilirubin/ALP/ALT

  * twice the upper limit of normal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Feasibility of the study | 18 months
  Time taken to recruit the required subjects (n=50)

SECONDARY OUTCOMES:
Clinical Outcomes | 6 months
  Death and hospitalisation rates
Clinical outcomes | 6 months
  Changes in office BP
Clinical outcomes | 6 months
  Changes in 6minute walk test
Clinical outcomes | 6 months
  Changes in echocardiographic left ventricular ejection fraction.

CONTACTS AND LOCATIONS:
Overall Officials: REGINA ASUKU, Study Director — CARDIOVASCULAR RESEARCH UNIT, UNIVERSITY OF ABUJA TEACHING HOSPITAL
Locations (1):
- University of Abuja Teaching Hospital, Abuja, Federal Capital Territory, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Sliwa K, et al. Readmission and death after an acute heart failure event: predictors and outcomes in sub-Saharan Africa: results from the THESUS-HF registry. Eur Heart J 2013; 34: 3151-59. 2. Cohn JN, et al. A randomized trial of the angiotensin-receptor blocker valsartan in chronic heart failure. N Engl J Med 2001; 345: 1667-75. 3. Lapu-Bula R, et al. From hypertension to heart failure: role of nitric oxide-mediated endothelial dysfunction and emerging insights from myocardial contrast echocardiography. Am J Cardiol 2007; 99: 7D-14D. 4. Taylor AL, et al. Combination of ISDN and hydralazine in blacks with heart failure. N Engl J Med 2004; 351: 2049-57. 5. Carson, P et al. Racial differences in response to therapy for heart failure: analysis of the vasodilator-heart failure trials. Vasodilator-Heart Failure Trial Study Group. J Card Fail 1999: 5; 178-87. 6. Damasceno A, et al. The causes, treatment, and outcome of acute heart failure in 1006 Africans from 9 countries. Arch Intern Med 2012; 172: 1386-94. 7. Sliwa K, et al. Bi treatment with hydralazine/nitrates vs. placebo in Africans admitted with acute HEart Failure (BA-HEF). Eur J Heart Fail 2016; 18: 1248-58.